CLINICAL TRIAL: NCT04160793
Title: Genital Nerve Stimulation - GNS - for Treatment of Non-neurogenic OAB
Acronym: GNS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prof. Dr. med. Marc Possover (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Marc Possover, Director, Possover International Medical Center AG
Organization: Possover International Medical Center AG (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GNS1
Record Dates: First submitted 2019-10-18; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Bladder, Overactive
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Prospective unblinded interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Genital Nerve Stimulation (Other): Stimulation of the DNP
  Interventions: Device: Genital Nerve Stimulation

INTERVENTIONS:
Device: Genital Nerve Stimulation — Implantation the vaginal way a stimulation's electrode to the dorsal nerve of the clintoris in local anesthesia

SUMMARY:
The Genital Nerve Stimulation - GNS - consists of a two-step procedure with a preoperative non-surgical test-phase and a final surgical implantation of the neuroprothesis. In contrast to the classical technique of transcutaneous lead electrode implantation for sacral or pudendal nerve stimulation, the GNS-test-phase does not require any interventional procedure: because the genital nerves are located just few millimeter below the skin, test-stimulation can be achieved using skin surface or needle electrodes. Stimulation is achieved using a battery powered hand-held stimulator . The effect of the stimulation can be tested by the patient in their daily, home and professional environment, or at the practice under urodynamic testing, or if required other electrophysio-logical testing. After confirmation of the effectiveness of GNS, implantation of a permanent neuroprothesis can be planned. The procedure is performed either under general or spinal anesthesia or using only local anesthesia with IV-sedation as in the classical tension-free vaginal tape procedure (TVT). Because the GNS does not require two surgical procedures for both the test- and the final-implantation but rather only one for the final implantation, the presented protocol allows considerable cost reduction in comparison to the usual procedures for sacral or pudendal nerve stimulation.

DETAILED DESCRIPTION:
Pelvic organ dysfunctions are complex and difficult to treat. These conditions affect a substantial portion of the population, especially with increasing age. The two most frequent pelvic dysfunctions are the idio-pathic overactive bladder (IOAB) and erectile dysfunction (ED).

In pelvic dysfunctions, sacral nerve stimulation was the first technique for pelvic nerves stimulation that typically involves electrical stimulation of the nerve via a dorsal transformational technique of implantation. SNS evolved as a widely used treatment for OAB but does not completely resolve symptoms in the majority of patients. Because PNS reach more "sphincter-vesico-anal" fibers than SNM, PNS has been proposed for patients who have failed to respond to sacral neuromodulation. The good effects of PNS in neurogenic and in some non-neurogenic disorders. However, the implantation of a lead to the PN is not easily accomplished and the risk for lead migration with implantation below the pelvic floor is increased. So there is definitively a need for a more suitable alternative for selective stimulation within the pelvic cavity, a method that cannot only be reserved for experts in this field but for all gynecologists dealing with patients suffering from functional disorders of the bladder in daily clinical practice. The stimulation of the dorsal nerve of the pe-nis/clitoris - GNS - emerges as a very attractive alternative that might result in great outcomes for controlling urinary and fecal disorders.

Because part of the DNP lies superficially to the skin outside the pelvis, this nerve can be stimulated using surface electrodes attached to the overlying skin of the penis or close to the clitoris. This application is however limited, due to intolerance to required high stimulation amplitude. Surface electrodes have limitations such as difficulties in proper daily placement and issues related to hygiene as well as a lack of acceptance in some patients. Implanted electrodes are more suitable. However, implanted electrodes in the penis or near the clitoris, must endure the mechanical stress of penile erections and external pressure, carrying the risk of the cable/electrode breaking or being dislocated.

The GNS consists of a two-step procedure with a preoperative non-surgical test-phase and a final surgical implantation of the neuroprothesis. In contrast to the classical technique of transcutaneous lead electrode implantation for sacral or pudendal nerve stimulation, the GNS-test-phase does not require any interventional procedure: because the genital nerves are located just few millimeter below the skin, test-stimulation can be achieved using skin surface or needle electrodes. Stimulation is achieved using a battery powered hand-held stimulator . The effect of the stimulation can be tested by the patient in their daily, home and professional environment, or at the practice under urodynamic testing, or if required other electro-physiological testing. After confirmation of the effectiveness of GNS, implantation of a permanent neuroprothesis can be planned. The procedure is performed either under general or spinal anesthesia or using only local anesthesia with IV-sedation as in the classical tension-free vaginal tape procedure (TVT). Because the GNS does not require two surgical procedures for both the test- and the final-implantation but rather only one for the final implantation, the presented protocol allows considerable cost reduction in comparison to the usual procedures for sacral or pudendal nerve stimulation.

ELIGIBILITY:
Inclusion Criteria:

* women >18y
* suffering form intractable iOAB
* proved iOAB by urodynamic testing
* non pregnant
* good health
* patients demanding for therapy of iOAB and willing taking part to the study
* >6-9 months from last therapy with botulinum toxine A

Exclusion Criteria:

* pregnancy
* patients affected by a neurogenic condition
* any health condition being a contraindication for the procedure

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of bladder voiding | 6 months
  Patient's report on frequency of micturition

SECONDARY OUTCOMES:
Safety of the GNS procedure | 6 months
  Record of all pre- and postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Marc Possover, PhD, MD, Principal Investigator — PIMC
Locations (1):
- Possover, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Farag FF, Martens FM, Rijkhoff NJ, Heesakkers JP. Dorsal genital nerve stimulation in patients with detrusor overactivity: a systematic review. Curr Urol Rep. 2012 Oct;13(5):385-8. doi: 10.1007/s11934-012-0273-x. PMID 22865209
- [Result] Martens FM, Heesakkers JP, Rijkhoff NJ. Surgical access for electrical stimulation of the pudendal and dorsal genital nerves in the overactive bladder: a review. J Urol. 2011 Sep;186(3):798-804. doi: 10.1016/j.juro.2011.02.2696. Epub 2011 Jul 23. PMID 21788054